CLINICAL TRIAL: NCT05911217
Title: An Open-label, Single-arm, Multicenter, Phase Ib Clinical Trial to Evaluate the Efficacy and Safety of CT041 Autologous CAR T Cell Injection After Adjuvant Chemotherapy in Subjects With Pancreatic Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of CT041 After Adjuvant Chemotherapy for Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT041-ST-05
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
Keywords: Adjuvant therapy; Pancreatic Cancer; Claudin18.2; CLDN18.2; CAR T cell
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-claudin18.2 chimeric antigen receptor T-cell therapy (Experimental): Experimental: anti-claudin18.2 chimeric antigen receptor T-cell therapy Phase 1b: Evaluate the efficacy and safety of CT041
  Interventions: Drug: CT041 autologous CAR T-cell injection

INTERVENTIONS:
Drug: CT041 autologous CAR T-cell injection — Treatment with anti-claudin18.2 chimeric antigen receptor T-cell infusion. Up to 3 times CT041 autologous CAR T-cell injection infusion
  Other Names: Single Group Assignment

SUMMARY:
An open-label, single-arm, multicenter, Phase Ib clinical trial to evaluate the efficacy and safety of CT041 Autologous CAR T Cell Injection after adjuvant chemotherapy in subjects with pancreatic cancer.

DETAILED DESCRIPTION:
This study is an open, multicenter, Phase Ib clinical trial evaluating chimeric antigen receptor-modified autologous T cells targeting Claudin18.2 (CLDN18.2) (CT041 autologous CAR T) in subjects with CLDN18.2 expression-positive pancreatic cancer who has undergone adjuvant chemotherapy. The aim of this study is to evaluate the efficacy, safety of CT041 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical trial; fully understand, be informed about this study and have signed the ICF; willing to follow and able to complete all study procedures;
2. Aged 18 to 79 years;
3. Histologically confirmed pancreatic ductal adenocarcinoma;
4. Macroscopic complete tumor removal (R0 or R1 resection);
5. Postoperative pathological stage (pTNM): T1-3, N0-2, M0;
6. Immunohistochemistry (IHC) staining of subject's tumor tissue sample is CLDN18.2-positive;
7. Subjects had recovered from surgery and had received 3 months of standard adjuvant therapy;
8. Abnormal CA19-9 level;
9. With sufficient venous access for leukapheresis collection;
10. ECOG performance status score 0-1;
11. Adequate organ function;
12. Men and women of childbearing potential must be willing to use effective methods of contraception to prevent pregnancy;

Exclusion Criteria:

1. Prior neoadjuvant therapy for pancreatic cancer;
2. Subjects with borderline resectable pancreatic cancer;
3. Present or past history of metastatic or locally recurrent pancreatic cancer;
4. Evidence of malignant ascites;
5. Subjects had diseases that may interfere with CA19-9 level, including but not limited to cholangitis, pancreatitis, obstructive jaundice, etc.
6. Toxicities caused by previous treatment have not recovered to CTCAE ≤ grade 2, except alopecia and other tolerable events as judged by the investigator or laboratory abnormalities allowed in this study;
7. Pregnant or lactating women;
8. Positive serology for HIV, Treponema pallidum or HCV;
9. Any active infections, including but not limited to active tuberculosis, HBV, EBV, CMV, COVID-19 infections;
10. Clinically significant thyroid dysfunction;
11. Previous allergy to immunotherapy and related drugs, allergy to CT041 ingredients and other serious allergic history;
12. Subjects who may be at high risk for potential digestive tract bleeding or perforation;
13. Known active autoimmune disease, including but not limited to, psoriasis or rheumatoid arthritis, or other conditions requiring long-term immunosuppressive therapy;
14. Subjects who have a history of organ transplantation or are awaiting organ transplantation;
15. Subjects who require anticoagulant therapy;
16. Subjects who are receiving or are expected to require long-term antiplatelet therapy during the study;
17. Subjects who have experienced major surgery or have significant trauma within 4 weeks before apheresis, or who are expected to undergo major surgery during the study period;
18. Previously received any gene-modified cell therapies (including CAR T, TCR T);
19. Subjects who have other serious diseases that may restrict them from participating in the study assessed by investigators;
20. Subjects with oxygen saturation ≤ 95%;
21. Subjects who have signs of central nervous system diseases or clinically significant neurological examination abnormalities;
22. Subjects who have other uncured malignant tumors in the past 3 years or at the same time, except those with very low degree of malignancy such as cervical cancer in situ and basal cell carcinoma of skin;
23. Vaccination with live attenuated vaccines within 4 weeks prior to apheresis or planned during the study;
24. Subjects who are unable to or unwilling to comply with the requirements of the study protocol as assessed by investigators.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Up to 18 months
  The time from the first infusion to the occurrence of local recurrence/distant metastasis or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs), treatment related AEs, AEs of special interest (AESI). | Up to 18 months
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
1 year DFS rate | Up to 18 months
  Proportion of patients alive without local recurrence/distant metastasis 1 year after the first infusion.
Metastasis free Survival (MFS) | Up to 18 months
  The time from the first infusion to the occurrence of any pancreatic cancer distant metastases or death from any cause, whichever occurred first.
Overall Survival (OS) | Up to 18 months
  The time from the first infusion to death of the subject from any cause.
The phamacokinetics in subjects receiving CT041 infusion in this study | Up to 18 months
  Peak cell expansion, peak expansion, area under the curve (AUC), and duration of cell survival after infusion of CT041 cells.
The immunogenicity in subjects receiving CT041 infusion in this study | Up to 18 months
  Drug antibody (ADA) positive rate after infusion of CT041 cells.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, Ph.D, Principal Investigator — Fudan University
Locations (8):
- China (8):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Hua zhong University of Science and Technology, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Ruijin Hospital, affiliated to Shanghai Jiaotong University, school of medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No